CLINICAL TRIAL: NCT03360409
Title: Compare Different Cervical Anterior Discectomy Procedures for Cervical Degenerative Disc Disease by After Procedure Sagittal Alignment on Radiograph :a Multiple Center Randomized Controlled Trial
Brief Title: Compare Different Cervical Anterior Discectomy Procedures by After Procedure Sagittal Alignment on Radiograph
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Zhenqi, department of spinal surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACD3
Record Dates: First submitted 2017-11-26; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Cervical Disc Degeneration
Keywords: Cervical Disc Degeneration; cervical anterior discectomy; Spinal alignment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- grade 1 (Experimental): ACD
  Interventions: Procedure: ACD
- grade 2 (Active Comparator): ACDF
  Interventions: Procedure: ACDF
- grade 3 (Active Comparator): ACDA
  Interventions: Procedure: ACDA

INTERVENTIONS:
Procedure: ACD — Undertake anterior cervical discectomy without fusion
  Arms: grade 1
Procedure: ACDF — anterior cervical discectomy with fusion
  Arms: grade 2
Procedure: ACDA — anterior cervical discectomy with arthroplasty
  Arms: grade 3

SUMMARY:
Patients with single-level cervical degenerative disc disease commonly undertook anterior discectomy. To compare the effect of anterior cervical discectomy without fusion (ACD), anterior cervical discectomy with fusion by stand-alone cage (ACDF) or anterior cervical discectomy with arthroplasty (ACDA)， a multiple center randomised controlled trial will be performed in patients with single-level cervical disease. The primary outcome will be cervical alignment by upright cervical spine radiographs estimated by Harrison posterior tangent method.

DETAILED DESCRIPTION:
This study will use a multiple center open-label randomised controlled trial to estimate the effect of ACD, ACDF, ACDA for single-level cervical degenerative disc. Patients with arm pain not responding to conservative treatment take part in this trial. They will be randomised assigned into 3 parallel arms. The participants in the each arm will undertake ACD ACDF or ACDA. The baseline is the day of surgery. The Harrison posterior tangent method was used as an estimate for measuring cervical alignment. The primary outcome will be the cervical sagittal alignment estimated by Harrison posterior tangent method.

ELIGIBILITY:
Inclusion Criteria:

* patients with arm pain not responding to conservative treatment
* lasted longer than 10 weeks
* single level disc degeneration
* mobile spine on dynamic lateral cervical X-rays

Exclusion Criteria:

* severe cardiopulmonary comorbidity
* suspected underlying malignant disease
* radicular syndrome
* spinal-cord compression syndrome
* contraindication for radiography

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
change of cervical alignment | 1 day postoperatively, 6 weeks, 3 months, 1 year and 2 years
  The Harrison posterior tangent method was used as an estimate for curvature

SECONDARY OUTCOMES:
quality of life | 1 day postoperatively, 6 weeks, 3 months, 1 year and 2 years
  Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO)

CONTACTS AND LOCATIONS:
Overall Officials: zhenqi zhu, Study Director — PekingUPH department of spinal surgery

IPD SHARING:
Plan to Share IPD: No